CLINICAL TRIAL: NCT01640262
Title: Evaluation of Modern MRI in the Diagnosis of Prostate Cancer in a Danish Setup
Status: Completed | Type: Observational
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Other Study IDs: H-1-2011-066
Record Dates: First submitted 2012-06-26; First posted 2012-07-13 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2014-05

CONDITIONS: Prostatic Neoplasms
Keywords: prostate biopsy; prostate cancer; Magnetic Resonance Imaging; Neoplasm Staging
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- localized prostate cancer: Danish men with localized prostate cancer
  Interventions: Other: Multiparametric magnetic resonance imaging (mMRI)

INTERVENTIONS:
Other: Multiparametric magnetic resonance imaging (mMRI) — A mMRI is performed before treatment of the patient and is compared to the standard diagnostic tools for evaluating the clinical stage and diagnose of prostate cancer

SUMMARY:
Clinical staging of prostate cancer in Denmark is determined solely by digital rectal examination and sometimes by TRUS, even though the investigators know these examinations are inaccurate and have limitations. Since the majority of men diagnosed with prostate cancer will die with their disease and not of their disease, and the different treatment-options may imply greater side effects, it is important to improve the diagnostic localization and staging of the tumour for optimal clinical management and therapy selection.

The development of modern multiparametric-high-field-magnetic-imaging (mMRI) offers new possibilities and approaches in detection, localization and staging of prostate cancer due to its high resolution and soft-tissue contrast. mMRI can provide information about the morphological, metabolic and cellular changes and characterize tissue- and tumour- vascularity and correlate it with tumour aggressiveness. This helps to locate and stage a possible tumour and to guide targeted-biopsies towards disease-suspicious areas. Internationally published data support the rapidly growing use of multiparametric MRI, as being the most sensitive and specific imaging tool for prostate cancer patients.

While mMRI internationally is a well recognized and accepted method for detection, localization and staging of prostate cancer, the use of mMRI in the diagnosis of PCa in Denmark has never been applied. Therefore, this project is carried out in order to evaluate the use of modern mMRI in the diagnosis of prostate cancer in a Danish setup.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is now the most frequently diagnosed male malignant disease in Denmark with more than 4000 new cases each year. PCa is the second leading cause of cancer related mortality in the western world. During their lifetime, one in six men will be clinically diagnosed with Prostate cancer and approximately one out of thirty will die of the disease. We know from autopsies that more than half of the male-population above the age of 60 is found to have histological cancer-changes. Therefore, the majority of men with histological proven cancer-changes will never develop a clinical disease that would affect their morbidity and mortality.

An elevated PSA (blood sample) and/or an abnormal rectal examination are indications of PCa. The diagnosis is made by trans-rectal-ultrasound guided biopsies (TRUS-biopsies) followed by histological examination. Each biopsy-session includes 10 to 12 biopsy-cores taken from standard locations throughout the prostate. Since over 40 % of the cancers are isoechoic on ultrasound and cannot be seen, there is a high risk that the tumour is either missed or that the most aggressive part of the tumour is not biopsied.

If you find a prostate cancer, it is important to know if the cancer is localized within the prostate or if it grows outside of the capsule. This is called staging and is essential in determine the best treatment-strategy and the patient's prognosis. In Denmark, staging is determined by digital rectal examination and sometimes by TRUS, even though we know these examinations are inaccurate and have limitations. It is important to improve the diagnostic localization and staging of the tumour for optimal clinical management and therapy selection.

The development of modern multiparametric-high-field-magnetic-imaging (mMRI) offers new possibilities and approaches in detection, localization and staging of prostate cancer due to its high resolution and soft-tissue contrast. mMRI can provide information about the morphological, metabolic and cellular changes and characterize tissue- and tumour- vascularity and correlate it with tumour aggressiveness. This helps to locate and stage a possible tumour and to guide targeted-biopsies towards disease-suspicious areas. Internationally published data support the rapidly growing use of multiparametric MRI, as being the most sensitive and specific imaging tool for prostate cancer patients.

The primary objective of this project is to investigate whether the use of modern MRI in Denmark can:

* Improve the diagnosis of Danish men suspected of prostate cancer and
* Improve the diagnosis and treatment planning of Danish men with biopsy-proven prostate cancer.

The secondary goal is to gain experience in the use of modern MRI in Denmark to evaluate prostatic tumors. This study forms the basis for investigating whether modern MRI should be used as an adjunct diagnostic tool for selected patients in the diagnosis of prostate cancer.

The project contains three separate studies evaluating the adjunct diagnostic value of mMRI to the conventional standard diagnostic evaluation and treatment.

The three studies:

* Study 1 is offered to patients with newly diagnosed localized non-metastatic prostate cancer and is comparing mMRI to TRUS and DRE in clinical classification of the cancer.
* Study 2 is offered to patients with newly diagnosed localized non-metastatic prostate cancer who underwent Brachytherapy and is comparing mMRI to CT-scan performed 4 weeks after surgery in the evaluation of postoperative dosimetry (treatment effect).
* Study 3 is offered to patients scheduled for re-biopsy due to continuing suspicion of prostate cancer after standard TRUS-guided biopsies with negative findings to see if multiparametric MRI can detect prostate cancer invisible on transrectal ultrasound; in order to improve detection rate.

ELIGIBILITY:
Inclusion Criteria Study 1:

* Patients with newly diagnosed localized (T1-2) or locally advanced (T3)prostate cancer

Exclusion Criteria Study 1:

* Metastatic prostate cancer
* Prostate cancer treatment
* Known allergic reaction to Gadolinium-based MRI contrast agent
* Prostate biopsy during the last 21 days
* Impaired renal function with GFR < 30 ml / min
* pacemaker
* Magnetic metal residues in the body
* Claustrophobia
* Psychiatric disorders
* Age under 18 years

Inclusion Criteria Study 2:

- Patients with localized prostate cancer who underwent brachytherapy 4 weeks prior to MRI.

Exclusion Criteria Study 2:

* Metastatic prostate cancer
* Prostate cancer treatment other than Brachytherapy
* Known allergic reaction to Gadolinium-based MRI contrast agent
* Prostate biopsy during the last 21 days
* Impaired renal function with GFR < 30 ml / min
* pacemaker
* Magnetic metal residues in the body
* Claustrophobia
* Psychiatric disorders
* Age under 18 years

Inclusion Criteria Study 3:

* Patients scheduled for re-biopsy due to continuing suspicion of prostate cancer after standard TRUS-guided biopsies with negative findings.

Exclusion Criteria Study 3:

* Histological positive prostate biopsies and known prostate cancer
* Metastatic prostate cancer
* Known allergic reaction to Gadolinium-based MRI contrast agent
* Prostate biopsy during the last 21 days
* Impaired renal function with GFR < 30 ml / min
* pacemaker
* Magnetic metal residues in the body
* Claustrophobia
* Psychiatric disorders
* Age under 18 years

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Study 1 is offered to 140 patients with newly diagnosed localized prostate cancer and is comparing mMRI to TRUS and DRE in the assessment of the clinical stage of prostate cancer.
  * Study 2 is offered to 55 patients with newly diagnosed localized prostate cancer who have undergone Brachytherapy and is comparing MRI to CT scan performed 4 weeks after surgery in the evaluation of postoperative dosimetry (treatment effect).
  * Study 3 is offered to 55 patients scheduled for re-biopsy due to continuing suspicion of prostate cancer after standard TRUS-guided biopsies with negative findings. Standardised TRUS-guided re-biopsies as well as TRUS biopsies of any MRI-suspicious lesion are performed in the same session and marked separately. The MRI-targeted biopsies are compared to the standard TRUS-guided re-biopsies to see if multiparametric MRI can detect prostate cancer invisible on transrectal ultrasound; in order to improve detection rate.
Sampling Method: Non-Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2011-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Change in the diagnosis and treatment planning based on MRI examination | The participants will be followed for the duration of the hospital diagnostic investagation, an expected average of 4 weeks
  Study 1: Change in clinical T-stage (TNM-classification) at baseline compared to the patological T-stage after curative treatment approx. 4 weeks later.
  Study 2: Change in prostatic volumen expressed in milliliter(ml) on CT and MRI 4 weeks after brachytherapy-operation compared to the prostatic volumen on TRUS at baseline.
  Study 3: Change detectionrate of prostatecancer using MRI-targeted biopsies.

SECONDARY OUTCOMES:
To gain experience in the use of modern multiparametric MRI in Denmark to evaluate prostatic tumors. | 2 years
  This study forms the basis for investigating whether modern MRI should be used as an adjunct diagnostic tool for selected patients in the diagnosis of prostate cancer

CONTACTS AND LOCATIONS:
Overall Officials: Lars P. Boesen, M.D., Principal Investigator — Department of Urology and Radiology
Locations (1):
- Department of Urology, Herlev University Hospital, Herlev, Herlev, Denmark